CLINICAL TRIAL: NCT03856554
Title: Comparison of Radiologic and Clinical Outcome of Single Level Lumbar Interbody Fusion Between Unilateral or Bilateral Facetectomy : Prospective Randomized Controlled Trial
Brief Title: Unilateral Versus Bilateral TLIF for Degenerative Lumbar Spondylolisthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Woo-Kie Min, Associate Professor, Spine Center and Department of Orthopedic Surgery, Kyungpook National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNUH 2017-04-021-004
Record Dates: First submitted 2018-03-07; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Degenerative Spondylolisthesis; Transforaminal Lumbar Interbody Fusion

STUDY DESIGN:
Intervention Model Description: Transforminal lumbar interbody fusion
  : unilateral versus bilateral facetectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients indicated for TLIF (Experimental): Patients with lumbar degenerative spondylolisthesis, indicated for TLIF surgery
  Interventions: Procedure: Unilateral Transforaminal Interbody fusion; Procedure: Bilateral Transforaminal Interbody fusion

INTERVENTIONS:
Procedure: Unilateral Transforaminal Interbody fusion — TLIF via unilateral factectomy and insertion of one cage
Procedure: Bilateral Transforaminal Interbody fusion — TLIF via bilateral factectomy and insertion of two cages

SUMMARY:
A prospective randomized controlled trial for comparison of radiologic outcomes of "single level transforaminal interbody fusion(TLIF) technique via unilateral versus bilateral facetectomy for the treatment of lumbar degenerative spondylolisthesis

DETAILED DESCRIPTION:
Traditionally many spine surgeons prefer single level TLIF surgery via bilateral facetectomy for increasing union rate. Our hypothesis - "Single level TLIF via unilateral facetectomy is sufficient for achieve successful fusion rate"

ELIGIBILITY:
Inclusion Criteria:

* lumbar degenerative spondylolisthesis
* indicated for surgery

Exclusion Criteria:

* not agreed for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Sagittal balance | through study completion, an average of 1 year
  Radiologic parameters
Interbody fusion(union) failure | through study completion, an average of 1 year
  Radiologic parameters. Use dynamic plain X-ray. Union defined as no movement at segment

SECONDARY OUTCOMES:
Pain scores | through study completion, an average of 1 year
  Visual analog scale
Functional scores | through study completion, an average of 1 year
  36-Item Short Form Survey (SF-36) Scoring

CONTACTS AND LOCATIONS:
Locations (1):
- Spine Center, Kyoungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No